CLINICAL TRIAL: NCT05108740
Title: Managed Access Program (MAP) Cohort Treatment Plan CRAD001Y2002M to Provide Access to Afinitor for Patients With Advanced Hormone Receptor Positive (HR+) Breast Cancer
Brief Title: MAP Treatment Plan With Afinitor for Postmenopausal Women With Advanced HR+ Breast Cancer
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRAD001Y2002M
Record Dates: First submitted 2021-09-09; First posted 2021-11-05 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Advanced Hormone Receptor Positive (HR+) Breast Cancer
Keywords: Breast Cancer; MAP; Hormone receptor positive; Afinitor; everolimus
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: everolimus — Self-administered as a daily dose of 10mg orally
  Other Names: Afinitor

SUMMARY:
The purpose of this Managed Access Program (MAP) Cohort Treatment Plan is to provide guidance to the Physician for the treatment and monitoring of patients in the Cohort MAP.

DETAILED DESCRIPTION:
Prior to inclusion of a patient in the Cohort, the requesting Physician must submit a request for access to the product in GEMS (Grants, External Requests and Managed Access System) accessible through https://www.novartis.com/our-focus/healthcare-professionals/managedaccess-programs providing the rationale for the request and relevant medical history of the patient.

The request is then assessed against the MAP and Cohort inclusion/exclusion criteria by the medical team experienced with the product and indication. Upon the required approvals, the patient is included in the Cohort.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this Treatment Plan have to meet all of the following criteria:

1. Patient has histological or cytological confirmation of hormone-receptor positive (HR+) breast cancer.
2. Patient is a postmenopausal woman: Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (i.e. age appropriate history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
3. Patient has recurrence or progression of their cancer after treatment with Femara® (letrozole) or Arimidex® (anastrozole).
4. Patient is willing to be treated with concomitant exemestane.
5. Patient has adequate bone marrow and coagulation function as shown by: absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L; platelets ≥ 100 × 10^9/L; hemoglobin (Hgb) ≥ 9.0 g/dL.
6. Patient has adequate liver function as shown by:

   * Total serum bilirubin ≤ 2.0 mg/dL,
   * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 ULN (or ≤ 5x ULN in patients with liver metastases),
   * INR ≤2.
7. Patient has adequate renal function as shown by serum creatinine ≤ 1.5 × ULN.
8. Patient has fasting serum cholesterol ≤ 300mg/dL or 7.75 mmol/L and fasting triglycerides ≤ 2.5 × ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
9. Patient will give a written informed consent obtained according to local guidelines.

Exclusion Criteria:

Patients eligible for this Treatment Plan must not meet any of the following criteria:

History of hypersensitivity to any drugs or metabolites of similar chemical classes as the product.

1. Patient has HER2- overexpression confirmed by local laboratory testing (IHC 3+ staining or in situ hybridization positive).
2. Patient requires chemotherapy for symptomatic visceral disease.
3. Patient is currently receiving hormone replacement therapy.
4. Patient has had prior therapy with mTOR inhibitors (e.g. sirolimus, temsirolimus, deforolimus).
5. Patient has a known intolerance or hypersensitivity to everolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus).
6. Patient is receiving treatment with systemic corticosteroids or other immunosuppressive agents.
7. Patient with a known history of HIV seropositivity.
8. Patient has uncontrolled diabetes as defined by fasting serum glucose >1.5× ULN despite adequate therapy. Patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout participation in the program and adjusted as necessary.
9. Patient has any severe and/or uncontrolled medical conditions such as:

   * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤6 months prior to randomization, serious uncontrolled cardiac arrhythmia,
   * Active or uncontrolled severe infection,
   * Liver disease such as cirrhosis, decompensated liver disease, and chronic hepatitis (i.e. quantifiable HBV-DNA and/or positive HbsAg, quantifiable HCV-RNA),
   * Known severely impaired lung function (spirometry and DLCO 50% or less of normal and O2 saturation 88% or less at rest on room air),
   * Active, bleeding diathesis.
10. Patient is unwilling to or unable to comply with the treatment plan.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal woman